CLINICAL TRIAL: NCT00385944
Title: A Randomized Double-Blind Cross-Over Study Comparing the Pharmacodynamic (PD)Response in Subjects With ACS Receiving 14 Days 10-mg Maintenance Dose (MD) Prasugrel vs 14 Days 150-mg MD Clopidogrel After Using a 900-mg Loading Dose (LD) of Clopidogrel to Reduce Ongoing Platelet Activation
Brief Title: The Effect on Blood Cells, Known as Platelets, Using Prasugrel vs Clopidogrel in Patients With the Heart Problem Acute Coronary Syndrome (ACS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10632; H7T-MC-TABN (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Experimental): Open label lead-in one time dose of Clopidogrel 900 mg oral tablets (a single or cumulative dose) and 250 mg to 500 mg aspirin loading dose (LD), either orally or intravenously. Patients are then assigned to maintenance dose (MD) prasugrel 10 mg and two placebo tablets, matched to clopidogrel, and 100 mg aspirin, all taken orally once a day for 14 days. Patients cross-over to MD of clopidogrel two 75 mg tablets and one placebo matched to prasugrel and 100 mg aspirin, all taken orally once a day for the next 14 days.
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Open label lead-in one time dose of Clopidogrel 900 mg oral tablets (a single or cumulative dose) and 250 mg to 500 mg aspirin loading dose (LD), either orally or intravenously. Patients are then assigned to maintenance dose (MD) Clopidogrel two 75 mg and one placebo tablet, matched to prasugrel, and 100 mg aspirin, all taken orally once a day for 14 days. Patients cross-over to MD of prasugrel one 10 mg tablet and two placebo tablets matched to clopidogrel and 100 mg aspirin, all taken orally once a day for the next 14 days.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10-mg tablet taken orally as a daily maintenance dose for a 14-day treatment period.
  Other Names: LY640315; Effient; Efient
  Arms: Prasugrel
Drug: Clopidogrel — Clopidogrel two 75-mg tablets taken orally as a daily maintenance dose for a 14-day treatment period.
  Arms: Clopidogrel

SUMMARY:
This is a multicenter, randomized, double-blind, cross-over study to compare the pharmacodynamic response in subjects with Acute Coronary Syndrome receiving a 10-mg maintenance dose (MD) of prasugrel compared with a 150-mg maintenance dose of clopidogrel, following a 900-mg loading dose (LD) of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Present with acute coronary syndrome (ACS) and have planned treatment with a one-time 900-mg loading dose of commercially available clopidogrel (administered as a single or cumulative dose).
* Are between the ages of 18 and 85 years.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Have overt ST-segment elevation myocardial infarction (STEMI).
* Have cardiogenic shock.
* Have refractory ventricular arrhythmias.
* Have New York Heart Association (NYHA) Class IV congestive heart failure.
* Have severe and uncontrolled hypertension.
* Have active internal bleeding or history of bleeding diathesis.
* Have an increased risk of bleeding.
* Have history of cerebrovascular accidents.
* Have certain abnormal blood level values.
* Are currently receiving chemotherapy or radiation therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 56 patients received a clopidogrel loading dose (LD) of 900 mg and were then randomized to receive a maintenance dose (MD) of either 10-mg prasugrel or 150-mg clopidogrel. Two patients withdrew from the study after randomization but prior to receiving a MD, one due to subject decision and one due to physician decision.
Groups:
- Prasugrel/Clopidogrel: One time oral loading dose (LD) of 900-mg clopidogrel (a single or cumulative dose)followed by a once daily MD of prasugrel 10 mg and 100 mg aspirin, for 14 days. Patients cross-over to a daily MD of clopidogrel 150 mg and 100 mg aspirin for an additional 14 days.
- Clopidogrel/Prasugrel: One time oral loading dose (LD) of 900-mg clopidogrel (a single or cumulative dose)followed by a once daily MD of clopidogrel 150 mg and 100 mg aspirin, for 14 days. Patients cross-over to a daily MD of prasugrel 10 mg and 100 mg aspirin for an additional 14 days.
- Loading Dose: Clopidogrel 900-mg Loading Dose (a single or cumulative dose)
Period: Loading Dose
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel | Loading Dose
Started | 0 | 0 | 56
Completed | 0 | 0 | 56
Not Completed | 0 | 0 | 0
Period: 1st Maintenance Dose Period
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel | Loading Dose
Started | 29 | 25 (Two patients withdrew from the study after randomization but prior to receiving the 1st MD.) | 0
Completed | 25 | 24 | 0
Not Completed | 4 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Entry Criteria Exclusion | 0 | 1 | 0
Not completed — Invalid Pharmacodynamic Data | 3 | 0 | 0
Period: 2nd Maintenance Dose Period
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel | Loading Dose
Started | 24 (1 patient discontinued prior to the 2nd MD Period (Sponsor decision due to early study termination)) | 22 (2 patients discontinued prior to the 2nd MD Period (Sponsor decision due to early study termination)) | 0
Completed | 22 | 19 | 0
Not Completed | 2 | 3 | 0
Not completed — Invalid PD Data | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel/Clopidogrel: One time oral loading dose (LD) of 900-mg clopidogrel (a single or cumulative dose) followed by a once daily MD of prasugrel 10 mg and 100 mg aspirin, for 14 days. Patients cross-over to a daily MD of clopidogrel 150 mg and 100 mg aspirin for an additional 14 days.
- Clopidogrel/Prasugrel: One time oral loading dose (LD) of 900-mg clopidogrel (a single or cumulative dose) followed by a once daily MD of clopidogrel 150 mg and 100 mg aspirin, for 14 days. Patients cross-over to a daily MD of prasugrel 10 mg and 100 mg aspirin for an additional 14 days.
- Total: Total of all reporting groups
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel | Total
Number analyzed (Participants) | 29 | 27 | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (13.7) | 58 (10.7) | 61 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 26 | 21 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 28 | 25 | 53
  African | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  France | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Maximum Platelet Aggregation (MPA) to 20 Micromolar (μM) Adenosine Diphosphate (ADP)
Description: Maximum platelet aggregation (MPA) to 20 μM adenosine diphosphate (ADP) was assessed by light transmission aggregometry (LTA).
Time Frame: 14 days after maintenance dose (MD)
Population: The primary analysis was performed on the intent-to-treat (ITT) population, that is, all randomized subjects with a maintenance dose MPA measured for at least one of the treatments.
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Groups:
- Prasugrel: Prasugrel (10-mg MD) + Aspirin (≤100-mg MD) (Prasugrel + Aspirin is administered once daily, either in the first or second MD period)
- Clopidogrel: Clopidogrel (150-mg MD) + Aspirin (≤100-mg MD) (Clopidogrel + Aspirin is administered once daily, either in the first or second MD periods)
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage aggregation | 27.1 (10.55) | 40.3 (14.96)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -12.91, 95% CI 2-sided [-17.02 to -8.81]

2. Secondary Outcome: MPA to 5 μM ADP
Description: Maximum platelet aggregation to 5 μM ADP was assessed by LTA.
Time Frame: 14 days after maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage aggregation | 16.9 (8.3) | 25.0 (11.09)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.81, 95% CI 2-sided [-10.96 to -4.65]

3. Secondary Outcome: Mean Residual Platelet Aggregation (RPA) to 20 µM ADP
Description: Residual platelet aggregation is the percentage (%) aggregation value as measured by LTA at 6 minutes after the addition of ADP.
Time Frame: 14 days after maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage aggregation | 9.4 (11.43) | 21.6 (21.54)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -11.98, 95% CI 2-sided [-17.06 to -6.90]

4. Secondary Outcome: Mean Residual Platelet Aggregation (RPA) to 5 µM ADP
Description: as for outcome 3
Time Frame: 14 days after maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage aggregation | 2.7 (5.26) | 7.1 (10.64)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -4.3, 95% CI 2-sided [-6.84 to -1.76]

5. Secondary Outcome: Inhibition Platelet Aggregation (IPA) to 20 μM ADP
Description: IPA is calculated as a percent decrease of MPA from baseline using the following formula:
  ([MPA at baseline - MPA at time of postbaseline] / MPA at baseline) x 100%
Time Frame: 14 days after maintenance dose (MD)
Population: Note: This was calculated only for subjects with a true clopidogrel-free measure at baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 22 | 21
Percentage inhibition | 64.2 (14.39) | 48.5 (18.58)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 15.16, 95% CI 2-sided [7.05 to 23.26]

6. Secondary Outcome: Inhibition Platelet Aggregation (IPA) to 5 μM ADP
Description: as for outcome 5
Time Frame: 14 days after maintenance dose (MD)
Population: Note: This was calculated only for subjects with a true clopidogrel-free measure at baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 22 | 21
Percentage inhibition | 72.4 (12.76) | 58.8 (17.33)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = 12.69, 95% CI 2-sided [5.56 to 19.81]

7. Secondary Outcome: Inhibition of Residual Platelet Aggregation (IRPA) to 20 μM ADP
Description: IRPA is calculated as a percent decrease of RPA from baseline using the following formula:
  ([RPA at baseline - RPA at time of postbaseline] / RPA at baseline) x 100%
Time Frame: 14 days after maintenance dose (MD)
Population: Note: This was calculated only for subjects with a true clopidogrel-free measure at baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 23 | 23
Percentage inhibition | 87.1 (15.26) | 75.9 (25.99)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; Mean Difference (Net) = 10.26, 95% CI 2-sided [2.17 to 18.34]

8. Secondary Outcome: Inhibition of Residual Platelet Aggregation (IRPA) to 5 μM ADP
Description: as for outcome 7
Time Frame: 14 days after maintenance dose (MD)
Population: Note: This was calculated only for subjects with a true clopidogrel-free measure at baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 23 | 23
Percentage inhibition | 95.6 (6.5) | 91.4 (15.18)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p = 0.123, Mixed Models Analysis; Mean Difference (Net) = 3.85, 95% CI 2-sided [-1.13 to 8.84]

9. Secondary Outcome: Platelet Reactivity Index (PRI)
Description: Platelet Reactivity Index percentage was assessed by Vasodilator-stimulated phosphoprotein (VASP). PRI percent (%) was calculated using the median fluorescence intensity (MFI) of samples included with prostaglandin E1 (PGE1) and ADP, according to the following formula:
  PRI%=[(MFI(PGE1)-MFI(PGE1 + ADP)/MFI(PGE1)]x100
  Lower PRI% values indicate greater P2Y12 receptor blockade.
Time Frame: 14 days after maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage PRI
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Percentage PRI | 22.1 (14.33) | 39.4 (21.05)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -16.83, 95% CI 2-sided [-23.05 to -10.62]

10. Secondary Outcome: P2Y12 Reaction Units (PRU)
Description: P2Y12 Reaction Units (PRU) assessed by Accumetrics Verify NowTM P2Y12. PRU represents the rate and extent of adenosine (ADP)-stimulated platelet aggregation. Lower values indicate greater P2Y12 platelet inhibition.
Time Frame: 14 days after maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 47 | 47
PRU | 44 (38.59) | 98.7 (63.69)
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -54.44, 95% CI 2-sided [-70.87 to -38.01]

11. Secondary Outcome: Poor Responder of MPA to 20 μM ADP Following Maintenance Dose (MD)
Description: Poor responder is defined as MPA to 20 μM ADP >75th percentile of the value at 6-18 hours post-clopidogrel LD.
Time Frame: 14 days after maintenance dose (MD)
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 49 | 47
Participants
  Responder | 48 | 35
  Poor Responder | 1 | 12

12. Secondary Outcome: Change in MPA to 20 μM ADP From Baseline to 6-18 Hrs Post Loading Dose (LD)
Description: Maximum platelet aggregation to 20 μM ADP was assessed by LTA.
Time Frame: Baseline to 6-18 hrs post loading dose (LD)
Population: Note: This was calculated only for subjects with a true clopidogrel-free measure at baseline (Visit 1)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Groups:
- Clopidogrel 900 mg: Clopidogrel 900 mg LD (a single or cumulative dose)
Arm/Group | Clopidogrel 900 mg
Number analyzed (Participants) | 23
Percentage aggregation | -35.5 (17.5)
Statistical Analysis 1: Comparison: Clopidogrel 900 mg; Test type: Superiority or Other; p < .001, two-sided paired t-test; Mean Difference (Net) = -35.5

13. Secondary Outcome: Change in MPA to 20 μM ADP From 6-18 Hrs Post Loading Dose (LD) to 14 Days After the First Maintenance Dose (MD)
Description: Maximum platelet aggregation to 20 μM ADP was assessed by LTA.
Time Frame: 6-18 hrs post loading dose (LD) to 14 days after the first maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Groups:
- Prasugrel/Clopidgrel: Prasugrel (10-mg MD) or Clopidogrel (150-mg MD) + Aspirin (≤100-mg MD)
- Clopidogrel/Prasugrel: Clopidogrel (150-mg MD)or Prasugrel (10-mg MD) + Aspirin (≤100-mg MD)
Arm/Group | Prasugrel/Clopidgrel | Clopidogrel/Prasugrel
Number analyzed (Participants) | 23 | 20
Percentage aggregation | -9 (15.71) | -0.6 (12.56)
Statistical Analysis 1: Comparison: Prasugrel/Clopidgrel; Paired t-test for each arm separately; Test type: Superiority or Other; p = 0.011, two-sided paired t-test; Mean Difference (Net) = -9
Statistical Analysis 2: Comparison: Clopidogrel/Prasugrel; Paired t-test for each arm separately; Test type: Superiority or Other; p = 0.847, two-sided paired t-test; Mean Difference (Net) = -0.6

14. Secondary Outcome: MPA to 20 μM ADP at 14 Days After the First Maintenance Dose (MD)
Description: Maximum platelet aggregation to 20 μM ADP was assessed by LTA.
Time Frame: 14 days after the first maintenance dose (MD)
Population: Subjects providing evaluable MPA to 20 μM ADP at 14 days after the first maintenance dose (MD)
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Groups:
- Prasugrel/Clopidogrel: Prasugrel (10-mg MD) or Clopidogrel (150-mg MD) + Aspirin (≤100-mg MD)
- Clopidogrel/Prasugrel: Clopidogrel (150-mg MD) or Prasugrel (10-mg MD) + Aspirin (≤100-mg MD)
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel
Number analyzed (Participants) | 27 | 24
Percentage aggregation | 28.9 (11.14) | 38.2 (12.86)
Statistical Analysis 1: Comparison: Prasugrel/Clopidogrel vs Clopidogrel/Prasugrel; Test type: Superiority or Other; p = 0.008, t-test, 2 sided; Mean Difference (Net) = -9.24, 95% CI 2-sided [-15.99 to -2.49]

15. Secondary Outcome: MPA to 20 μM ADP at 14 Days After the Second Maintenance Dose (MD)
Description: Maximum platelet aggregation to 20 μM ADP was assessed by LTA.
Time Frame: 14 days after the second maintenance dose (MD)
Population: Subjects providing evaluable MPA to 20 μM ADP at Day 29.
Measure: Mean (Standard Deviation); unit: Percentage aggregation
Arm/Group | Prasugrel/Clopidogrel | Clopidogrel/Prasugrel
Number analyzed (Participants) | 23 | 22
Percentage aggregation | 42.5 (16.89) | 25 (9.58)
Statistical Analysis 1: Comparison: Prasugrel/Clopidogrel vs Clopidogrel/Prasugrel; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Median Difference (Net) = 17.52, 95% CI 2-sided [9.22 to 25.83]

16. Secondary Outcome: Number of Participants With Bleeding Events According to Thrombolysis in Myocardial Infarction Study Group (TIMI) Criteria
Description: Bleeding events will be classified as Major Bleeding, Minor Bleeding, or Insignificant Bleeding according to the TIMI criteria. Major bleeding: any intracranial hemorrhage (ICH) OR any clinically overt bleeding (including bleeding evident on imaging studies) associated with a fall in hemoglobin (Hgb) of ≥5 gm/dL from baseline. Minor Bleeding: any clinically overt bleeding associated with a fall in Hgb of ≥3 grams/deciliter (gm/dL) but <5 gm/dL from baseline. Insignificant bleeding: any bleeding event that does not meet criteria for a Major or Minor bleed.
Time Frame: 14 days after maintenance dose (MD)
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 51 | 49
Participants
  Major | 0 | 0
  Minor | 0 | 1
  Insignificant | 3 | 1

17. Secondary Outcome: Number of Participants With Bleeding Events According to Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO)
Description: Bleeding events will be classified according to the GUSTO definitions as follows: Severe or Life-Threatening Bleeding: any ICH OR any bleeding event resulting in substantial hemodynamic compromise requiring treatment. Moderate Bleeding: any bleeding event resulting in the need for transfusion. Minor bleeding: any other bleeding event that does not require transfusion or cause hemodynamic compromise.
Time Frame: 14 days after maintenance dose (MD)
Measure: Number; unit: Participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 51 | 49
Participants
  Severe or life-threatening | 0 | 0
  Moderate | 0 | 0
  Minor | 3 | 2

18. Secondary Outcome: Correlation of MPA to 20 μM ADP and PRU
Description: Pearson-correlation estimated between MPA to 20 μM ADP and Accumetrics VerifyNowTM P2Y12 PRU
Time Frame: Baseline through 29 days of treatment
Measure: Number; unit: Correlation coefficient
Groups:
- Intent-to-treat Population: Both clopidogrel and prasugrel combined population
Arm/Group | Intent-to-treat Population
Number analyzed (Participants) | 56
Correlation coefficient | 0.8

ADVERSE EVENTS:
Groups:
- Clopidogrel 900 mg LD: One time oral loading dose (LD) of 900-mg clopidogrel
- Prasugrel 10 mg - 1st MD: Once daily MD of prasugrel 10 mg and 100 mg aspirin, for 14 days.
- Clopidogrel 150 mg - 1st MD: Once daily MD of clopidogrel 150 mg and 100 mg aspirin, for 14 days.
- Clopidogrel 150 mg - Crossover From Prasugrel 10 mg: Once daily MD of clopidogrel 150 mg and 100 mg aspirin, for an additional 14 days. These are patients who received a daily MD of prasugrel 10 mg and 100 mg aspirin during the 1st MD period.
- Prasugrel 10 mg - Crossover From Clopidogrel 150 mg: Once daily MD of prasugrel 10 mg and 100 mg aspirin, for an additional 14 days. These are patients who received a daily MD of clopidogrel 150 mg and 100 mg aspirin during the 1st MD period.
Arm/Group | Clopidogrel 900 mg LD | Prasugrel 10 mg - 1st MD | Clopidogrel 150 mg - 1st MD | Clopidogrel 150 mg - Crossover From Prasugrel 10 mg | Prasugrel 10 mg - Crossover From Clopidogrel 150 mg
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/29 | 0/25 | 1/24 | 1/22
Other Adverse Events (participants affected / at risk) | 20/56 | 7/29 | 7/25 | 3/24 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 900 mg LD (N=56) | Prasugrel 10 mg - 1st MD (N=29) | Clopidogrel 150 mg - 1st MD (N=25) | Clopidogrel 150 mg - Crossover From Prasugrel 10 mg (N=24) | Prasugrel 10 mg - Crossover From Clopidogrel 150 mg (N=22)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 900 mg LD (N=56) | Prasugrel 10 mg - 1st MD (N=29) | Clopidogrel 150 mg - 1st MD (N=25) | Clopidogrel 150 mg - Crossover From Prasugrel 10 mg (N=24) | Prasugrel 10 mg - Crossover From Clopidogrel 150 mg (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days